CLINICAL TRIAL: NCT00054158
Title: A Phase II Study of VAD (Vincristine, Adriamycin, Dexamethasone) Plus Thalidomide (Low Dose) as Frontline Therapy for Newly Diagnosed Patients With Multiple Myeloma (MM)
Brief Title: Combination Chemotherapy and Thalidomide in Treating Patients With Stage I, Stage II, or Stage III Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Masking: None | Purpose: Treatment
Other Study IDs: RP 02-15; RPCI-RP-0215
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Dexamethasone; Doxorubicin; Thalidomide; Vincristine

INTERVENTIONS:
Drug: dexamethasone
Drug: doxorubicin hydrochloride
Drug: thalidomide
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Thalidomide may stop the growth of cancer by stopping blood flow to the tumor. Combining chemotherapy with thalidomide may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and thalidomide in treating patients who have newly diagnosed stage I, stage II, or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall response rate in patients with newly diagnosed stage I, II, or III multiple myeloma treated with vincristine, doxorubicin, dexamethasone, and low-dose thalidomide.
* Determine the ability to collect peripheral blood stem cells in patients after treatment with this regimen.

OUTLINE: This is an open-label, nonrandomized study.

Patients receive vincristine IV and doxorubicin IV continuously on days 1-4 and oral dexamethasone on days 1-4, 9-12, and 17-20. Patients also receive low-dose oral thalidomide daily on days 1-28. Treatment repeats every 4 weeks for 4-6 courses in the absence of disease progression.

Patients are followed until disease progression or bone marrow transplantation.

PROJECTED ACCRUAL: Approximately 17-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed stage I, II, or III multiple myeloma (MM)
* No refractory or relapsed MM

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin less than 1.5 mg/dL
* AST less than 2.5 times upper limit of normal

Renal

* Not specified

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 effective methods of contraception (including at least 1 highly active method) for at least 4 weeks before, during, and for at least 4 weeks after study participation
* No active serious infections uncontrolled by antibiotics
* No insufficient mental capacity that would preclude informed consent
* No other medical condition or reason that would preclude study participation
* Willing and able to comply with the FDA-mandated S.T.E.P.S program

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior thalidomide

Chemotherapy

* No more than 1 course of prior vincristine, doxorubicin, and dexamethasone

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent alcohol consumption

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher A. Chanan-Khan, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States